CLINICAL TRIAL: NCT00335634
Title: Sexual Dysfunction and Adaptation in Couples Affected by Prostate Cancer Surgery: Steps Towards a Bio-Psychosocial Model of Treatment
Brief Title: Sexual Dysfunction and Adaptation in Couples Affected by Prostate Cancer Surgery
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: PC-05-0813
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer; Erectile Dysfunction Following Radical Prostatectomy; Sexual Dysfunction
Keywords: Prostate Cancer; Radical Prostatectomy; Sexual Dysfunction; Intimacy; Adaptation; Psychosocial Oncology
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to explore patient and partner experiences with sexual dysfunction following radical prostatectomy, in order to understand its effects on sexual and non-sexual intimacy. This will enable us to provide assistance in the future to individuals experiencing similar circumstances.

DETAILED DESCRIPTION:
We are studying the impact of sexual dysfunction following radical prostatectomy on patient and partners' experiences of intimacy. Research with men in post-radical prostatectomy recovery indicates 25%-75% experience sexual dysfunction. Many patients experience anxiety and distress related to sexual difficulties. These experiences may progress and result in long-term problems in the relationship between patients and their partners. Despite apparent levels of effectiveness, up to half of the patients who turn to sexually assistive aids after surgical removal of the prostate discontinue use of the aids within one year. Additionally, difficulties in communicating about sexual impairments can significantly interfere with the couples' ability to achieve successful adaptation. We are interested in studying patient and partner experiences with sexual dysfunction in order to understand its effects on sexual and non-sexual intimacy.

Participation in this study will involve completing 6 confidential face-to-face interviews on three separate occasions (3-6 months, 12-15 months, and 21-24 months post-surgery). On each occasion, participants will be required to take part in a "couple's" interview with his/her partner, as well as an individual interview. The interviews will provide participants with the opportunity to discuss the impact of sexual dysfunction on mood, thoughts, and communication with their partners. Demographic information will be collected at the initial interview. As well, at each of the 3 time points, participants will also be asked to complete a questionnaire package containing 6 psychological questionnaires. All questionnaires and interview material will be kept strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* Radical prostatectomy treatment for prostate cancer at Princess Margaret Hospital or Etobicoke General Hospital
* At least 3 months, but less than 6 months post-radical prostatectomy
* Experience sexual dysfunction as a result of radical prostatectomy
* Must have an intimate partner and be able to participate as a couple

Exclusion Criteria:

* Detectable prostate specific antigen (PSA) post-radical prostatectomy
* Patient or partner unable to speak English
* Patient or partner unwilling to allow interviews to be recorded
* Patient or partner unwilling to participate

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer who have had a radical prostatectomy, and their intimate partners.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Semi-Structured Interview - Patient | 3-6 months post-radical prostatectomy
Semi-Structured Interview - Patient | 12-15 months post-radical prostatectomy
Semi-Structured Interview - Patient | 21-24 months post-radical prostatectomy
Semi-Structured Interview - Partner | 3-6 months post-radical prostatectomy
Semi-Structured Interview - Partner | 12-15 months post-radical prostatectomy
Semi-Structured Interview - Partner | 21-24 months post-radical prostatectomy
Semi-Structured Interview - Couple | 3-6 months post-radical prostatectomy
Semi-Structured Interview - Couple | 12-15 months post-radical prostatectomy
Semi-Structured Interview - Couple | 21-24 months post-radical prostatectomy

SECONDARY OUTCOMES:
The International Index of Erectile Function | 3-6 months post-radical prostatectomy
  Used to assess erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall sexual satisfaction in patients and male partners
Index of Sexual Life | 3-6 months post-radical prostatectomy
  Used to assess sexual desire and overall sexual satisfaction in female partners
Dyadic Adjustment Scale | 3-6 months post-radical prostatectomy
  Used to measure couple distress
Hospital Anxiety and Depression Scale | 3-6 months post-radical prostatectomy
  Used to measure anxiety and depression
The International Index of Erectile Function | 12-15 months post-radical prostatectomy
  Used to assess erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall sexual satisfaction in patients and male partners
The International Index of Erectile Function | 21-24 months post-radical prostatectomy
  Used to assess erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall sexual satisfaction in patients and male partners
Index of Sexual Life | 12-15 months post-radical prostatectomy
  Used to assess sexual desire and overall sexual satisfaction in female partners
Index of Sexual Life | 21-24 months post-radical prostatectomy
  Used to assess sexual desire and overall sexual satisfaction in female partners
Dyadic Adjustment Scale | 12-15 months post-radical prostatectomy
  Used to measure couple distress
Dyadic Adjustment Scale | 21-24 months post-radical prostatectomy
  Used to measure couple distress
Hospital Anxiety and Depression Scale | 12-15 months post-radical prostatectomy
  Used to measure anxiety and depression
Hospital Anxiety and Depression Scale | 21-24 months post-radical prostatectomy
  Used to measure anxiety and depression
Brief Profile of Mood States | 3-6 months post-radical prostatectomy
  Used to measure emotional distress
Brief Profile of Mood States | 12-15 months post-radical prostatectomy
  Used to measure emotional distress
Brief Profile of Mood States | 21-24 months post-radical prostatectomy
  Used to measure emotional distress
Miller Social Intimacy Scale | 3-6 months post-radical prostatectomy
  Used to measure patient-partner intimacy
Miller Social Intimacy Scale | 12-15 months post-radical prostatectomy
  Used to measure patient-partner intimacy
Miller Social Intimacy Scale | 21-24 months post-radical prostatectomy
  Used to measure patient-partner intimacy
Sternberg Triangular Love Scale | 3-6 months post-radical prostatectomy
  Used to assess levels of intimacy (closeness and connectedness), commitment and decisions to love, and passion
Sternberg Triangular Love Scale | 12-15 months post-radical prostatectomy
  Used to assess levels of intimacy (closeness and connectedness), commitment and decisions to love, and passion
Sternberg Triangular Love Scale | 21-24 months post-radical prostatectomy
  Used to assess levels of intimacy (closeness and connectedness), commitment and decisions to love, and passion

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Matthew, PhD, C.Psych, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Etobicoke General Hospital, Etobicoke, Ontario
  - The Prostate Centre, Princess Margaret Hospital, Toronto, Ontario